CLINICAL TRIAL: NCT00582777
Title: African American Study of Kidney Disease and Hypertension ABPM Pilot Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Lawrence Agodoa, M.D., NIDDK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AASK ABPM Pilot (completed); 7 U01 KD04868
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Hypertensive Renal Disease
Keywords: nocturnal blood pressure; chronic renal disease; hypertensive renal disease; African Americans; ABPM
MeSH Terms: conditions — Hypertensive Nephropathy; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- USUAL (Active Comparator): USUAL treatment - The patient's antihypertensive regimen at the baseline visit is the comparison (or control) regimen. All once a day medications will be administered in the morning.
  Interventions: Behavioral: USUAL - take your BP Meds as you usually do
- HS Dosing (Experimental): HS DOSING - In this period, the patient's antihypertensive regimen at the baseline visit will be standardized for the once/day medications to be given at bedtime.
  * For those on monotherapy with a once/day antihypertensive regimen, the time of administration will be changed to bed time.
  * For those on multi-drug therapy, the time of administration of all once a day antihypertensive drugs will be changed to bed time.
  Interventions: Behavioral: HS DOSING
- ADD-ON DOSING (Experimental): ADD-ON DOSING - This regimen will start with the USUAL regimen to which an additional agent will be added at bed time. An additional dose of ramipril, diltiazem, or hydralazine are three possible options for the add on medication. The intent of the ADD ON therapy is to lower nocturnal BP with minimal impact on daytime BP. Thus, agents with < 24 hr duration of action are preferred. The specific choice and dose of add-on therapy (of the three agents) will be up to the site investigator considering the clinical situation of each participant based on the guidelines below.
  Interventions: Drug: ADD On Dosing

INTERVENTIONS:
Behavioral: USUAL - take your BP Meds as you usually do — The patient's antihypertensive regimen at the baseline visit is the comparison (or control) regimen. All once a day medications will be administered in the morning.
  Arms: USUAL
Behavioral: HS DOSING — Take your usual BP meds at bed time
  Arms: HS Dosing
Drug: ADD On Dosing — Take your usual BP meds but add one more med at bed time.
  Arms: ADD-ON DOSING

SUMMARY:
4. Methods 4a. Overview The study will be conducted in participants in the African-American Study of Kidney Disease (AASK) Cohort study as a randomized three period cross-over trial.

Eighty five percent of AASK cohort participants are currently on an ACE inhibitor or angiotensin receptor blocker; the most commonly used ACE inhibitor is ramipril. The new strategies proposed in this pilot study will remain ramipril-based, to maintain the overall blood pressure control achieved thus far.

The antihypertensive regimens proposed are as follows:

* AM dosing of ramipril and other once daily medications in the participants antihypertensive regimen (termed USUAL),
* Bedtime dosing of ramipril and other once a day medications in the participant's antihypertensive regimen (termed HS-DOSING), and
* their current antihypertensive regimen plus an additional antihypertensive agent dosed at bed time; the choice of the additional agent will be tailored based on prespecified clinical guidelines (termed ADD-ON DOSING)

The "usual arm" serves as the comparator arm. The "hs dosing" and "add-on dosing" arms test practical strategies that could be tested in a subsequent clinical outcomes trial and that could be implemented in clinical practice. We hypothesize that both arms will reduce nocturnal BP in comparison to "usual dosing". We further hypothesize that the "hs dosing" arm will raise daytime BP somewhat but have no net effect on 24 hour BP and that the "add on dosing" arm will have no effect on daytime BP but lower 24 hour BP.

This pilot study will begin after the last scheduled AASK Cohort study visit. Eligible participants will be treated for 6 weeks on each of 3 antihypertensive regimens. The sequence of the regimens will be random. Each period of the three periods will have 2 visits, one visit at 3 weeks and one visit at 6 weeks. In the last week of each 6-week period, a 24-hour ABPM will be obtained. The primary outcome variable is nocturnal BP; each pair wise difference between the regimens will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the AASK Cohort Study
* Ability and willingness to provide informed consent
* Completion of a technically adequate ABPM at CO48 AASK cohort study visit.
* Participants must have had at least 2 visits in the last 12 months of the Cohort Study (July 1 2006 to June 1 2007)
* The average of last two BPs measured at least one week apart in the Cohort Study must be less than or equal to 140/90 mm Hg. This would exclude a small percentage of the AASK cohort population; however, it would enroll a group of participants with stable BP who should not require adjustments to their antihypertensive medications during the course of this study.
* Antihypertensive medications at baseline visit: This refers to the participant's antihypertensive regimen at the time of the baseline visit ; the transition period may be used to adjust the participant's antihypertensive regimen to meet these criteria, based on the clinical judgement of the site investigator.

Exclusion Criteria:

* Arm circumference greater than 50 cms.
* ESRD requiring renal replacement therapy or kidney transplantation
* Institutionalized participants
* Shift workers working at night
* MI or CVA within 3 months of AASK Cohort close out visit
* Participants with known ejection fraction less than 40%
* Females known to be pregnant or lactating
* Participants likely to reach end stage renal disease within the next six weeks, in the judgement of the site investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Night Time Blood Pressure | Night time blood pressure from APBM at weeks 6, 12, and 18

SECONDARY OUTCOMES:
Blood pressure in the clinic Daytime blood pressure | Measured at weeks 6, 12, and 18

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, M.D., Study Chair — University Hospitals, Cleveland; Jackson T. Wright, Jr., MD, Ph.D., FACP, Principal Investigator — University Hospitals Cleveland Medical Center; Janice Lea, MD, Principal Investigator — Emory Center for Hypertension and Renal Disease Research; Francis B. Gabbai, MD, Principal Investigator — University of Calirfornia, San Diego; Otelio S. Randall, MD, Principal Investigator — Howard University; Lawrence Appel, MD, MPH, Principal Investigator — Johns Hopkins University; Keith Norris, MD, Principal Investigator — Charles Drew Medical Center; DeAnna Cheek, MD, Principal Investigator — Medical University of South Carolina; Michael Lipkowitz, MD, Principal Investigator — Lenox Hill Hospital; Lee Hebert, MD, Principal Investigator — Ohio State University; George Bakris, MD, Principal Investigator — University of Chicago; Stephen G. Rostand, MD, Principal Investigator — University of Alabama at Birmingham; Geraldine Bichier, MD, Principal Investigator — University of Florida; Gabriel Contreras, MD, Principal Investigator — University of Miami; Kenneth Jamerson, MD, Principal Investigator — University of Michigan; Miroslav J. Smogorzewski, MD, Principal Investigator — University of Southern California; Robert D. Toto, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Julia A. Lewis, MD, Principal Investigator — Vanderbilt University
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Charles Drew Medical College, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Lenox Hill Hospital, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Univesity of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Juraschek SP, Appel LJ, Miller ER 3rd. Metoprolol Increases Uric Acid and Risk of Gout in African Americans With Chronic Kidney Disease Attributed to Hypertension. Am J Hypertens. 2017 Sep 1;30(9):871-875. doi: 10.1093/ajh/hpx113. PMID 28830083
- [Derived] Rahman M, Greene T, Phillips RA, Agodoa LY, Bakris GL, Charleston J, Contreras G, Gabbai F, Hiremath L, Jamerson K, Kendrick C, Kusek JW, Lash JP, Lea J, Miller ER 3rd, Rostand S, Toto R, Wang X, Wright JT Jr, Appel LJ. A trial of 2 strategies to reduce nocturnal blood pressure in blacks with chronic kidney disease. Hypertension. 2013 Jan;61(1):82-8. doi: 10.1161/HYPERTENSIONAHA.112.200477. Epub 2012 Nov 19. PMID 23172931